CLINICAL TRIAL: NCT01105403
Title: A Phase IIa, Proof of Concept Study is to Determine the Degree of Mobilisation of CD34+ Cells Following Administration of POL6326 in Patients With Multiple Myeloma
Brief Title: Exploratory Study on POL6326 in Stem Cell Mobilization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Polyphor Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POL-2
Record Dates: First submitted 2010-04-13; First posted 2010-04-16 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Multiple Myeloma
Keywords: Hematopoietic stem cells; Mobilisation; Autologous transplantation
MeSH Terms: conditions — Multiple Myeloma | interventions — balixafortide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CD34+ mobilisation for transplantation (Experimental)
  Interventions: Drug: POL6326

INTERVENTIONS:
Drug: POL6326 — IV infusion of POL6326 followed by apheresis to collect mobilized stem cells from peripheral blood
  Other Names: not appicable

SUMMARY:
The purpose of this study is to determine whether POL6326 is safe and clinically active to mobilize hematopoietic stem cells followed by transplantation

ELIGIBILITY:
Inclusion Criteria:

1. Have multiple myeloma in Stage II or III, according to the criteria of Durie and Salmon.
2. Male or female between 18 and 70 years of age, inclusive. Male and females capable of reproduction must agree to use adequate contraceptive measures (e.g. condom, intrauterine device, oral contraceptive) until 3 months after termination of treatment.
3. Measurable disease, defined by one of the following:

   * Serum M protein ≥1.0 g/dL by protein electrophoresis
   * Quantifiable immunoglobulin levels and/or
   * urinary M protein excretion ≥200 mg/24 hours.
4. All patients have undergone 3 cycles of chemotherapy, with the last dose of chemotherapy given 3 to 8 weeks before study entry.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 2.
6. Life expectancy of >6 months.
7. Have given their written informed consent to participate in the study

Exclusion Criteria:

1. Have non-secretory myeloma and/or plasma cell leukaemia.
2. History of other malignancies during the past 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin, cervical carcinoma, or localised prostate carcinoma.
3. Any other clinically significant medical conditions.
4. History of cardiac disease NHYA classification ≥3.
5. Insufficient bone marrow, liver and renal function as assessed by the following clinical laboratory evaluations:

   Haemoglobin <9.0 g/L. Absolute neutrophil count <1500/µL. Platelet count <50000/µL. Total bilirubin >1.5 x upper limit of normal (ULN). Alanine aminotransferase (ALT) and alkaline phosphatase (AP) >2.5 x ULN. Amylase and lipase >1.5 x ULN. Serum creatinine >2.0 x ULN. Prothrombin time (PT) and activated partial thrombo-plastin time (aPTT) >1.5 x ULN.
6. Pregnant or lactating female patients.
7. Known history of HIV infection or chronic hepatitis B or C infection.
8. Receipt of immunotherapy, radiation therapy, or any investigational drug within 30 days of study drug administration.
9. Prior radiotherapy to more than 3 vertebrae.
10. Active serious bacterial or fungal infections; >grade 3 National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).
11. Receipt of haematopoietic cytokines within 10 days of study drug administration.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-04; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To assess the ability of POL6326 to mobilise CD34+ hematopoietic stem cells in patients with primary multiple myeloma | Up to four days
  Number of patients achieving the minimal number of CD34+ cells (≥2 x 10 mill/kg BW) collected during one to four cycles of apheresis which are considered necessary and safe to proceed with autotransplantation
  Number of apheresis cycles required to obtain the minimal number of CD34+ cells necessary for autotransplantation (≥2 x 10 mill/kg BW)

SECONDARY OUTCOMES:
To evaluate the safety and pharmacokinetics of POL6326 in patients with multiple myeloma | 2 months
To determine the efficacy of POL6326 in reconstitution of immune system after transplantation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Goldschmidt, MD, Principal Investigator — Heidelberg University
Locations (1):
- Department of Internal Medicine V, Heidelberg, Germany